CLINICAL TRIAL: NCT06200688
Title: The Effect of Peanut Ball Application on the Delivery Process, Birth Pain, and Birth Process: a Randomized Controlled Study
Brief Title: The Effect of Peanut Ball Application on Delivery Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, YELİZ YILDIRIM VARIŞOĞLU, Prof. Asist., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 745044
Record Dates: First submitted 2023-12-16; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Birth, First

STUDY DESIGN:
Intervention Model Description: Experimental Group: Pregnant women who received the peanut ball application were provided with necessary information about the ball and how to use it through visual aids showing the positions provided by the midwife. A total of 5 positions were shown to the pregnant women. The peanut ball was used when the cervical dilation reached 6 cm. Pregnant women in active labor, the transition phase, and the second stage with the peanut ball were directed to change positions every 30-45 minutes. Emphasis was placed on selecting positions in which the pregnant women felt comfortable.
  Control Group: No intervention was made other than routine practices within the clinic for pregnant women. It was observed that pregnant women generally spent the time before delivery lying down and connected to electronic fetal monitoring.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Ball Group (Experimental): In this group, pregnant women changed positions with a peanut ball during labor.
  Interventions: Other: PEANUT BALL
- Control Group (No Intervention): No intervention was applied in this group.

INTERVENTIONS:
Other: PEANUT BALL — Experimental Group: Pregnant women who were applied with a peanut ball were informed about the necessary information related to the ball by the midwife with a visual representation of the positions. A total of 5 positions were shown to the pregnant women. Peanut ball was started to be used when the cervical dilation reached 6 cm. Pregnant women in the active phase, the transition phase, and the second stage of labor where the peanut ball was applied were directed to change positions every 30-45 minutes. Importance was given to selecting positions where the pregnant woman felt comfortable.
  Control Group: No intervention was made other than routine practices within the clinic for pregnant women. It was generally observed that pregnant women spent the time until delivery lying down and connected to electronic fetal monitoring.
  Arms: Peanut Ball Group

SUMMARY:
This study was carried out to evaluate the effect of peanut ball application on labor process, birth pain, and birth comfort. The data of the study were collected between July 2021 and July 2022 in a Training and Research Hospital in Istanbul. 115 pregnant women who met the inclusion criteria of the study were included in the sampling, and the study was completed with 102 (experimental n: 51; control n: 51) pregnant women. Data were collected with an introductory information form, visual and verbal pain scales, Birth Comfort Scale, and birth follow-up form.

DETAILED DESCRIPTION:
A group was determined to be involved in the study after obtaining consent from the pregnant women participating in the research. The purpose of the study was explained to all pregnant women, informing them that the data would be anonymized and privacy principles would be adhered to.

Experimental Group: Pregnant women who received the peanut ball application were provided with necessary information about the ball and how to use it through visual aids showing the positions provided by the midwife. A total of 5 positions were shown to the pregnant women. The peanut ball was used when the cervical dilation reached 6 cm. Pregnant women in active labor, the transition phase, and the second stage with the peanut ball were directed to change positions every 30-45 minutes. Emphasis was placed on selecting positions in which the pregnant women felt comfortable.

Control Group: No intervention was made other than routine practices within the clinic for pregnant women. It was observed that pregnant women generally spent the time before delivery lying down and connected to electronic fetal monitoring.

In the Birth Monitoring Form, the gestational week found in the patient's file, interventions and medications applied in the first stage of labor, the situation of episiotomy application in the second stage, the newborn's birth time, and 1st and 5th APGAR scores, newborn's length, weight, head circumference, and gender were recorded. In both groups, labor pains during the dilation stage were evaluated three times using the Visual Anolog Scale (VAS) when the dilation was at 6 cm, 9 cm, and 10 cm. During this period, the pregnant women were asked to rate the pain they felt on the VAS scale from 1 to 10, and the values expressed were recorded by the researcher. The childbirth comfort scale and the form indicating mothers' views

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women
* 37w-40w gestational week (term)
* Pregnant women over the age of 18 years

Exclusion Criteria:

* Pregnant women who gave birth by cesarean section
* who had received epidural anesthesia/analgesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 102 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Birth duration | 1 day
  Birth duration was assessed using a partograph.
Birth pain | 8 hours
  Labor pains in the dilatation phase: dilation 6 cm, 9 cm and 10 cm with VAS It was evaluated 3 times in total during the time it was cm. During this period, pregnant women were asked to VAS They were asked to score the pain they felt between 1 and 10, and the expressed values were recorded by the researcher.
Birth comfort | 15 minutes
  The birth comfort scale was administered to pregnant women by the researcher within the first 4 hours after birth.

SECONDARY OUTCOMES:
Pregnancy introductory information | 15 minutes
  A pregnancy information form was used for all pregnant women after randomization to identify and evaluate the sociodemographic and socioeconomic information of the pregnant women.
Birth Follow-up | 1 day
  In the Birth Follow-up Form, it is included in the hospitalization file of the pregnant woman.
  gestational week, interventions and medications administered in the first stage of labor, Episiotomy application status in the second stage, newborn birth time, 1st and 5th APGAR and Newborn height, weight, head circumference and gender were evaluated and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: YELİZ YILDIRIM VARIŞOĞLU, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No